CLINICAL TRIAL: NCT03350451
Title: A Phase 2, Multicenter, Open-Label, Extension Study to Evaluate the Long-Term Administration of ALN-GO1 in Patients With Primary Hyperoxaluria Type 1
Brief Title: An Extension Study of an Investigational Drug, Lumasiran (ALN-GO1), in Participants With Primary Hyperoxaluria Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-GO1-002; 2016-003134-24 (EudraCT Number)
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: PH1; Primary Hyperoxaluria; RNAi Therapeutic; siRNA; AGT
Keywords: Hyperoxaluria, Primary; Hyperoxaluria; Kidney Diseases; Urologic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Metabolic Diseases
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria; Kidney Diseases; Urologic Diseases; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Metabolic Diseases | interventions — lumasiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M (Experimental): Participants enrolling from study 001B (NCT02706886), received lumasiran, subcutaneous (SC) injection, at a starting dose of 1.0 milligrams per kilograms (mg/kg) once monthly (QM) or 3.0 mg/kg once every 3 months [Q3M]) from Day 1 up to a maximum of Month 6. By Month 6, all participants were approved to change dose and/or dosing regimen to receive lumasiran, SC injection at a dose of 3.0 mg/kg, Q3M, up to Month 51 of the treatment period.
  All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6. As the cumulative dose administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the Safety Review Committee (SRC).
  Interventions: Drug: Lumasiran
- Lumasiran (ALN-GO1): 3.0 mg/kg QM (Experimental): Participants enrolling from study 001B, received lumasiran, SC injection, at a starting dose of 3.0 mg/kg, QM, from Day 1 up to a maximum of Month 21. By Month 21, all participants were approved to change dosing regimen to receive lumasiran, SC injection, at a dose of 3.0 mg/kg, Q3M, up to Month 51 of the treatment period.
  Interventions: Drug: Lumasiran

INTERVENTIONS:
Drug: Lumasiran — Multiple doses of lumasiran by SC injection
  Other Names: ALN-GO1

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of lumasiran in participants with Primary Hyperoxaluria Type 1.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 12 months of completion of Study ALN-GO1-001
* In the opinion of the investigator tolerated the study drug
* If taking Vitamin B6 (pyridoxine), willing to remain on a stable regimen for the study duration
* Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must be willing to use a highly effective method of contraception
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Clinically significant health concerns (with the exception of PH1)
* Clinically significant cardiovascular abnormality
* Abnormal for AST/ALT and any other clinical safety laboratory result considered clinically significant
* Requirement for chronic dialysis

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (9):
- France (3):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Paris
- Clinical Trial Site, Bonn, Germany
- Israel (2):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
- Clinical Trial Site, Amsterdam, Netherlands
- United Kingdom (2):
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 study centers in France, Germany, Israel, Netherlands and the United Kingdom from 04 April 2018 to 07 February 2023. A total of 20 participants previously treated in Study 001B (NCT02706886) were enrolled and treated in this study.
Pre-assignment Details: The cumulative dose of lumasiran administered over 6 months was the same for both 1 mg/kg once monthly (QM) & 3 mg/kg once every 3 months (Q3M), these participants were pooled into one arm as recommended by the Safety Review Committee (SRC). As pre-specified in the SAP, participants who began treatment at 1 mg/kg QM, then transitioned to 3 mg/kg Q3M were to be summarized as a single group. All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6.
Groups:
- Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M: Participants enrolling from study 001B, received lumasiran, subcutaneous (SC) injection, at a starting dose of 1.0 milligrams per kilograms (mg/kg) QM or 3.0 mg/kg (Q3M) from Day 1 up to a maximum of Month 6. By Month 6, all participants were approved to change dose and/or dosing regimen to receive lumasiran, SC injection at a dose of 3.0 mg/kg, Q3M, up to Month 51 of the treatment period.
  All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6. As the cumulative dose administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the SRC.
Period: Overall Study
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
Started | 13 | 7
Safety Analysis Set (Safety analysis set included all participants who received any amount of study drug.) | 13 | 7
Pharmacodynamic Analysis Set (Pharmacodynamic (PD) analysis set included all participants who received any amount of study drug and who had at least 1 post-dose urine sample for PD.) | 13 | 7
Completed | 13 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set. The cumulative dose of lumasiran administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the SRC. As pre-specified in the SAP, participants who began treatment at 1 mg/kg QM, then transitioned to 3 mg/kg Q3M were to be summarized as a single group. All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6.
Groups:
- Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M: Participants enrolling from study 001B, received lumasiran, SC injection, at a starting dose of 1.0 mg/kg QM or 3.0 mg/kg Q3M from Day 1 up to a maximum of Month 6. By Month 6, all participants were approved to change dose and/or dosing regimen to receive lumasiran, SC injection at a dose of 3.0 mg/kg, Q3M, up to Month 51 of the treatment period.
  All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6. As the cumulative dose administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the SRC.
- Total: Total of all reporting groups
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (12.31) | 12.6 (3.95) | 14.9 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 4
  White | 10 | 5 | 15
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: AE is any untoward medical occurrence in a participant or clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Safety analysis set included all participants who received any amount of study drug.
Time Frame: Baseline (Day -1) up to 54 months
Population: The cumulative dose of lumasiran administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the SRC. As pre-specified in the SAP, participants who began treatment at 1 mg/kg QM, then transitioned to 3 mg/kg Q3M were to be summarized as a single group. All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
Number analyzed (Participants) | 13 | 7
Participants | 13 | 7

2. Secondary Outcome: Change From Baseline in 24-hour Urinary Oxalate Corrected for Body Surface Area (BSA) at 54 Months
Description: Oxalate produced by the liver is the key toxic metabolite that drives disease pathology in participants with primary hyperoxaluria type 1 (PH1). The risk of disease complications increase continuously as oxalate levels increase. 24-hour urinary oxalate (millimole [mmol]/ 24 hour [h]/1.73 meters squared [m^2]) corrected for BSA at each visit per participant was calculated as follows: [Urine oxalate concentration (micromole per liter [umol/L])/1000 (umol/mmol)]*[24hour urine volume (mL)/1000 (mL/L)]* [24 hours/actual collection hours]*1.73/(BSA). Baseline was the derived baseline value from the lumasiran treated period of Study ALN-GO1-001. A negative change from baseline indicated a favorable outcome. PD analysis set included all participants who received any amount of study drug and who had at least 1 post-dose urine sample for PD. Overall number of participants analyzed are the number of participants with data available for analysis.
Time Frame: Baseline (Day -1) up to 54 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/24hr/1.73m^2
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
Number analyzed (Participants) | 12 | 6
mmol/24hr/1.73m^2 | -1.425 (0.2188) | -2.126 (0.5528)

3. Secondary Outcome: Change From Baseline in 24-hour Urinary Oxalate:Creatinine Ratio at 54 Months
Description: Baseline is the derived baseline value from the lumasiran treated period of Study ALN-GO1-001. A negative change from baseline indicates a favorable outcome. PD analysis set included all participants who received any amount of study drug and who had at least 1 post-dose urine sample for PD.
Time Frame: Baseline (Day -1) up to 54 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/mmol
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
Number analyzed (Participants) | 13 | 7
mmol/mmol | -0.2175 (0.03880) | -0.2480 (0.04047)

4. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at 54 Months
Description: Baseline was defined as the last measurement prior to the first dose of lumasiran in the ALN-GO1-001 study. eGFR was calculated based on the Modification of Diet in Renal Disease (MDRD) formula for participants >=18 years of age at enrollment and the Schwartz Bedside formula for participants <18 years of age at enrollment. eGFR based on MDRD formula was calculated as follows: eGFR (mL/min/1.73 m^2) = 175 × (serum creatinine {SCr} [μmol/deciliter(dL)]/88.4)-1.154 × (age)-0.203 × (0.742, if female), or × (1.212, if African American) and based on Schwartz formula: eGFR (mL/min/1.73m2) = (36.2 × height [cm])/ SCr (μmol /dL). Safety analysis set included all participants who received any amount of study drug.
Time Frame: Baseline (Day -1) up to 54 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
Number analyzed (Participants) | 13 | 7
mL/min/1.73m^2 | 0.674 (3.7970) | -12.026 (3.6369)

ADVERSE EVENTS:
Time Frame: Baseline (Day -1) up to 54 months
Description: Safety analysis set. The cumulative dose of lumasiran administered over 6 months was the same for both 1 mg/kg QM & 3 mg/kg Q3M, these participants were pooled into one arm as recommended by the SRC. As pre-specified in the SAP, participants who began treatment at 1 mg/kg QM, then transitioned to 3 mg/kg Q3M were to be summarized as a single group. All 3 participants who began treatment at 1 mg/kg QM transitioned to 3 mg/kg Q3M regimen by Month 6.
Arm/Group | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M | Lumasiran (ALN-GO1): 3.0 mg/kg QM
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/13 | 3/7
Other Adverse Events (participants affected / at risk) | 13/13 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M (N=13) | Lumasiran (ALN-GO1): 3.0 mg/kg QM (N=7)
Thyroid Mass (Endocrine disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Bone Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 1
Renal Stone Removal (Surgical and medical procedures) | 1 | 0
Thyroid Operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumasiran (ALN-GO1): 1.0 mg/kg QM or 3.0 mg/kg Q3M (N=13) | Lumasiran (ALN-GO1): 3.0 mg/kg QM (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Thyroid Mass (Endocrine disorders) | 0 | 1
Eye Allergy (Eye disorders) | 1 | 0
Periorbital Swelling (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 0 | 1
Feeling Cold (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 4 | 4
Non-cardiac Chest Pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Vaccination Site Pain (General disorders) | 1 | 1
Vessel Puncture Site Haematoma (General disorders) | 1 | 0
Immunisation Reaction (Immune system disorders) | 1 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 6 | 3
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cystitis Escherichia (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1
Tinea Versicolour (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb Injury (Injury, poisoning and procedural complications) | 2 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skin Wound (Injury, poisoning and procedural complications) | 1 | 0
Stoma Site Pain (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Bilirubin Conjugated Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 3 | 0
Blood Creatinine Increased (Investigations) | 0 | 1
Electrocardiogram QRS Complex Prolonged (Investigations) | 1 | 0
Glycolic Acid Increased (Investigations) | 0 | 1
SARS-CoV-2 Test Positive (Investigations) | 3 | 0
Ultrasound Breast Abnormal (Investigations) | 1 | 0
Ultrasound Kidney Abnormal (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 3
Weight Gain Poor (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 1
Device Breakage (Product Issues) | 0 | 1
Affective Disorder (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Sleep Disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal Cyst (Renal and urinary disorders) | 0 | 1
Renal Pain (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Genital Pain (Reproductive system and breast disorders) | 1 | 0
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy Closure (Surgical and medical procedures) | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 1
Wisdom Teeth Removal (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT03350451/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03350451/SAP_001.pdf